CLINICAL TRIAL: NCT02428816
Title: Evaluation and Validation of a Multimodal MRI Neuroimaging Method: Application to Differential Diagnosis and Disease Progression in Parkinsonian Syndromes
Brief Title: Evaluation of a Multimodal Neuroimaging Method for Diagnosis in Parkinsonian Syndromes
Acronym: MultiPAMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: C12-52; 2012-A01252-41 (Registry Identifier: IDRCB)
Record Dates: First submitted 2013-01-28; First posted 2015-04-29 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Parkinson's Disease; Multiple System Atrophy
Keywords: differential diagnosis; multimodal MRI; Parkinson's Disease; Multiple System Atrophy
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patients with Parkinson's Disease (Experimental): Patients with PD will be submitted to an MRI acquisition and to behavioural evaluations in each visits (two visits planned)
  Interventions: Other: MRI acquisition; Behavioral: behavioral evaluations
- Patients with MSA (Experimental): Patients with MSA will be submitted to an MRI acquisition and to behavioural evaluations in each visits (two visits planned)
  Interventions: Other: MRI acquisition; Behavioral: behavioral evaluations
- Controls (Experimental): 30 healthy controls will be submitted to an MRI acquisition and to behavioural evaluations in a sole visit
  Interventions: Other: MRI acquisition; Behavioral: behavioral evaluations

INTERVENTIONS:
Other: MRI acquisition — MRI acquisitions
Behavioral: behavioral evaluations — Evaluations about motor abilities, sleep, cognition and lifestyle

SUMMARY:
Based on previous promising results, the next step for the validation of a multimodal MRI method in diagnosis and follow up of patients reached by parkinsonian syndromes is (i) to test whether the multimodal neuroimaging is able to discriminate at the individual level, patients with multiple system atrophy parkinsonism (MSA) and patients with idiopathic Parkinson's disease (PD) (ii) to determine whether the method is sensitive to measure changes over time for the two diseases, according to imaging, neuropsychological and other clinical data. Patients will be compared with healthy controls.

DETAILED DESCRIPTION:
30 patients with PD, 30 patients with MSA and 30 healthy controls will be examined in a 3Tesla MRI.

The aim of our project is to demonstrate that our multimodal MRI method can discriminate both diseases with a similar clinical presentation and monitor the progress of the disease. CIC's expertise in recruitment and assessment of patients, and the powers of the INSERM U825 in terms of development and processing in neuroimaging guarantee the feasibility of the project and its successful completion.

ELIGIBILITY:
Inclusion Criteria:

* informed consent signed
* right handed patients
* Mini Mental Score > 22
* no other neurological disease than Parkinson's Disease (PD) or Multiple System Atrophy (MSA)
* non-demented patients reached by PD or MSA (according to diagnosis criteria from UK PD Brain Bank and from Gilman and colleagues, 1998, for PD and MSA respectively)
* for PD patients only : Hoehn and Yahr score from 2 to 3

Exclusion Criteria:

* claustrophobia
* contraindications to MRI (cardiac or auditive prothesis, pacemakers, cerebral clip, stimulating electrodes)
* pregnant women
* major neuropsychiatric disease
* refusal to be informed in case of cerebral anomaly detected during MRI acquisition
* uncompensated thyroid deficit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2013-01-24 (Actual); Primary Completion 2016-07-28 (Actual); Study Completion 2016-07-28 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure to discriminate individual patients and patients with MPI and AMS through multimodal MRI isolating multiparametric spatial signature resulting from a combination of markers in multimodal imaging. | 1 year

SECONDARY OUTCOMES:
correlate MP and MSA disease severity with extracted multimodal MRI biomarkers in whole brain | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Rascol, Pr, Principal Investigator — INSERM UMR 825, France
Locations (1):
- Inserm Umr 825, Toulouse, France